CLINICAL TRIAL: NCT03689088
Title: A Prospective Pilot Study Investigating the Use of a Sensing Contact Lens-based Device for 24-hour Monitoring of Intraocular Pressure in Healthy Subjects and Patients With Open Angle Glaucoma
Brief Title: Sensing Contact Lens-based Device for 24-hour Monitoring of Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: GF-1703
Record Dates: First submitted 2018-09-21; First posted 2018-09-28 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Glaucoma, Open-Angle; Healthy
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Manometry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational device (Goldfish) (Experimental): IOP will be monitored for 24 h in the Goldfish eye
  Interventions: Device: Goldfish
- Tonometry (Active Comparator): IOP will be acquired by standard tonometry at specific times in the the fellow eye
  Interventions: Device: Tonometry

INTERVENTIONS:
Device: Goldfish — Goldfish will be placed in the eye for 24h monitoring
  Arms: Investigational device (Goldfish)
Device: Tonometry — Fellow eye will be measured by tonometry
  Arms: Tonometry

SUMMARY:
Glaucoma is characterized by irreversible vision loss through the progressive death of optic nerve fibers unless timely diagnosis and adequate treatment are provided. Medical therapy is aimed at lowering intraocular pressure (IOP) below a clinically determined target level in order to prevent or slow glaucoma progression. IOP is known to vary with the time of day as well as with daily activities.

The current way of assessing nycthemeral IOP fluctuation is to perform repeated discrete tonometry measurements, allowing only snapshot and non-continuous measurements once per hour in the best cases. The procedure is cumbersome, expensive, inconvenient (disturbed sleep cycle as patient is awoken for nocturnal/sleep period measurements) and may not detect crucial IOP values in time.

Sensimed AG has developed a new contact lens (CL)-based device intended to continuously measure IOP over 24 hours. The objective of this study is to investigate the use of device for 24-hour IOP monitoring in healthy subjects and glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* For Open Angle Glaucoma (OAG) subjects, a clinical diagnosis of primary OAG, including normal tension glaucoma (NTG) all known untreated IOP measurements < 22 mmHg using Goldmann Applanation Tonometry (GAT) for NTG no IOP-lowering treatment; otherwise, a 4-week wash-out period prior to the recording
* For healthy subjects, no structural defects, normal visual fields, IOP ≤ 21 mmHg and open angles on gonioscopy
* Aged ≥ 18 years, either gender
* Body Mass Index ≤ 30 kg/m2
* Central Corneal Radius (flat meridian) between 7.5 mm (45 D) and 7.9 mm (42.75 D)
* Central Corneal Thickness between 500 microns and 600 microns
* Difference in IOP absolute value between eyes within 2.5 mmHg at screening in sitting position
* Same direction of IOP variation (positive or negative) for the 2 eyes when moving from sitting to supine positions at screening
* Spherical refraction within ±6.00 diopters and cylinder refraction within ±3.00 diopters
* Having given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Ocular pathology (other than glaucoma for glaucoma subjects)
* Previous glaucoma, cataract or refractive surgery
* Corneal or conjunctival abnormality, precluding contact lens adaptation
* Severe dry eye syndrome
* Subjects with allergy to corneal anesthetic
* Subjects with contraindications for silicone CL wear
* Subjects with contraindications for Water Drinking Test (WDT) (eg., heart, renal problems)
* Subjects unable or unwilling to comply with the study procedures
* Participation in other interventional clinical research within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Changes in IOP assessed by Goldfish following known physiological and induced changes in IOP | 24 hours
  IOP will be measured using tonometry in the fellow eye and compared to IOP measured in the Goldfish eye with the Goldfish device

SECONDARY OUTCOMES:
Percentage of subjects completing 24-hour session with Goldfish | 24 hours
  Percentage of subject completing the session will be calculated at the end of the study
Wearing discomfort of Goldfish based on visual analogue scale | 24 hours
  Tolerability of the Goldfish lens will be subjectively evaluated before and after GF wear using a visual analogue scale from 0 (no discomfort) to 100 (severe discomfort) mm
Evaluation of Goldfish technical performance based on the percentage of valid Goldfish measurements | 24 hours
  Percentage of valid measurement will be calculated at the end of each monitoring session
Correlation between IOP and ocular pulse amplitude (OPA) assessed by Goldfish in the Goldfish eye and IOP and OPA measured by tonometry in the fellow eye | 24 hours
  OPA will be extracted from the Goldfish signal in the Goldfish eye and measured by tonometry in the fellow eye. Both IOP and OPA measurement will be compared between fellow eyes
Relationship between Goldfish IOP and blood pressure (BP) measurements over 24 hours | 24 hours
  IOP signal acquired with Goldfish will be compared to BP signal assessed with a BP holter

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wasilewicz, MD, Principal Investigator — [W]-Eye Clinic
Locations (1):
- [W]-Eye clinic, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No